CLINICAL TRIAL: NCT03825484
Title: Expanded Access Program (EAP) for Patients With Advanced Cancers and FGFR Genetic Alterations Who Have Exhausted All Treatment Options
Brief Title: Expanded Access Program (EAP) for Participants With Advanced Cancers and Fibroblast Growth Factor Receptor (FGFR) Genetic Alterations Who Have Exhausted All Treatment Options
Status: Approved for marketing | Type: Expanded Access
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108489; 42756493MAF4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Advanced Cancers and FGFR Genetic Alterations
MeSH Terms: interventions — erdafitinib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Erdafitinib — Participants will start erdafitinib 8 milligram (mg) (formulated as tablets with 3 mg, 4 mg and 5 mg dosages) orally once daily until disease progression, intolerable toxicity, withdrawal of consent or decision by the doctor to discontinue treatment. Dose will be up-titrated to 9 mg based on serum phosphate levels and if there is no drug-related toxicity.
  Other Names: JNJ-42756493

SUMMARY:
The purpose of this program is to provide participants an early access to erdafitinib prior to market authorization (that is, Food and Drug Administration [FDA] approval in the United States). The program is limited to participants with advanced cancers and fibroblast growth factor receptor (FGFR) genetic alterations who have exhausted at least 2 lines of standard of care therapy and who are not eligible for an erdafitinib clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a documented fibroblast growth factor receptor (FGFR) alteration
* Participant does not have co-morbidities that would alter risk-benefit of providing erdafitinib (determined by treating physician's assessment)
* Life expectancy is greater than (>) 3 months (determined by treating physician's assessment)
* Participant has exhausted treatment options for their disease (review of prior treatments)
* Participant is not eligible for other erdafitinib clinical trials including but not limited to BLC3001/NCT03390504 and BLC2002/NCT03473743

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC